CLINICAL TRIAL: NCT03352063
Title: Effect of Prolonged Sitting on Metabolic and Cardiovascular Responses to Short-Term Exercise Training
Brief Title: Prolonged Sitting on Responses to Short-Term Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Edward F. Coyle, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-07-0074
Record Dates: First submitted 2017-10-09; First posted 2017-11-24 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Atherosclerosis; Metabolic Syndrome
MeSH Terms: conditions — Atherosclerosis; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either the sitting plus exercise or walking plus exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting with Exercise (Active Comparator): Subjects will complete a short term training protocol while sitting >11 hours per day. This training will be preceded by a VO2max test to aid in setting the correct intensity for training. Subjects will be asked to complete three high fat tolerance tests. One to establish a baseline, the second to determine the acute effects of training, and a third at the completion of training to determine the cumulative effect of exercise training.
  Interventions: Behavioral: Prolonged sitting with exercise
- Walking with exercise (Active Comparator): Subjects will complete a short term training protocol while sitting <5 hours per day. This training will be preceded by a VO2max test to aid in setting the correct intensity for training. Subjects will be asked to complete three high fat tolerance tests. One to establish a baseline, the second to determine the acute effects of training, and a third at the completion of training to determine the cumulative effect of exercise training.
  Interventions: Behavioral: Active walking with exercise.

INTERVENTIONS:
Behavioral: Prolonged sitting with exercise — Subjects will commit to sitting more than 11 hours per day and taking less than 5000 steps per day while participating in exercise training.
  Arms: Sitting with Exercise
Behavioral: Active walking with exercise. — Subjects will commit to sitting less than 5 hours per day and taking more than 10000 steps per day while participating in exercise training.
  Arms: Walking with exercise

SUMMARY:
Prolonged sitting has been shown to effect the response to a high fat tolerance test (HFTT) after acute exercise. This study will evaluate the effect of prolonged sitting on response to a HFTT after a short term training period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years

Exclusion Criteria:

* cardiovascular problems (e.g. pre-existing heart issues, coronary artery disease, hypertension, etc.)
* respiratory problems
* musculoskeletal problems that prevent prolonged sitting or exercise
* obesity
* susceptibility to fainting
* pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Plasma Triglycerides | 6 hours
  Areas under the curve for triglyceride concentration will be calculated for hourly samples from a 6-hour lipid tolerance test

SECONDARY OUTCOMES:
Plasma Insulin | 6 hours
  Areas under the curve for insulin concentration will be calculated for hourly samples from a 6-hour lipid tolerance test
Plasma glucose | 6 hours
  Areas under the curve for glucose concentration will be calculated for hourly samples from a 6-hour lipid tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton HM, Wolfe AS, Vardarli E, Satiroglu R, Coyle EF. Background Inactivity Blunts Metabolic Adaptations to Intense Short-Term Training. Med Sci Sports Exerc. 2021 Sep 1;53(9):1937-1944. doi: 10.1249/MSS.0000000000002646. PMID 34398061